CLINICAL TRIAL: NCT00226889
Title: Treatment of Early Systemic Sclerosis by Bosentan
Acronym: TRANOS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: failure of recruiting a sufficient number of patients
Sponsor: Rikshospitalet University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACTNR.2004-000650-23
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2006-03

CONDITIONS: Systemic Sclerosis (Scleroderma)
Keywords: Scleroderma; Fibrosis; Therapy; Bosentan; Endothelin-1
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Fibrosis | interventions — Bosentan

INTERVENTIONS:
Drug: bosentan

SUMMARY:
Systemic sclerosis (ssc) is characterised by extensive tissue fibrosis. Using drugs that are capable of inhibiting fibroblast activity may be beneficial if administrered early in the disease course. Thirty adult patients with early SSc will be treated with the endothelin-1 antagonist bosentan for 6 months.Disease progression will be assessed.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is characterised by obliterative vasculopathy and extensive fibrosis. The accumulation of extracellular components in the extracellular matrix is mostly due to increased activity og tissue fibroblasts. The proliferation and hyperactivity of the fibroblasts may be caused by enhanced production of several cytokins, among them endothelin-1.The activity of endothelin-1 has been shown to be increased both in the circulation and within skin lesions. Endothelin-1 has several distinct properties, among them profibrotic activity, inflammatory and vasoconstriction.Thus, the actions induced by endothelin-1 may be a potensial target for the therapy of SSc.

Thirty patients with early SSc, that is of less than 12 months duration will be offered six months of treatment with the oral dual endothelin-1 antagonist bosentan. Assessment of disease progression will be performed at 3, 6, 9. 12 and 24 months using clinical, histological and immunohistochemical methods.

ELIGIBILITY:
Inclusion Criteria:

* Early systemic sclerosis

Exclusion Criteria:

* Age > 70 or < 18
* Pregnancy
* Nursing
* HIV
* Hb < 8.5 g/l
* Systolic blood pressure < 85 mmHg
* Lack of compliance
* Liver disease
* Hypersensitivity to bosentan
* Concurrent us of glibenclamide, ciclosporine A or tacrolimus -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-01; Primary Completion 2009-01; Study Completion 2009-06

PRIMARY OUTCOMES:
Overall clinical progression
Degree of deposition of ET-1 in skin

SECONDARY OUTCOMES:
Development of extradermatological manifestations
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jan T Gran, Professor, Study Director — department of rheumatology
Locations (1):
- Department of rheumatology, Rikshospitalet, Oslo, Norway